CLINICAL TRIAL: NCT06952166
Title: Understanding the Psychological Benefits and Neurophysiological Mechanisms of Qigong in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15104721-2
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Qigong
MeSH Terms: interventions — Qigong; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Qigong (Baduanjin) (Experimental): 12-week training of Baduanjin, with two sessions per week. Each session lasts for 60 min.
  Interventions: Behavioral: Qigong (Baduanjin)
- Mindfulness-based intervention (Active Comparator): 12-week training of mindfulness-based breathing, walking, and stretching practices, with two sessions per week. Each session lasts for 60 min.
  Interventions: Behavioral: Mindfulness-based intervention
- Physical exercise (Active Comparator): 12-week training of stretching, flexibility exercise, and balance exercise, with two sessions per week. Each session lasts for 60 min.
  Interventions: Behavioral: Physical exercise
- Waitlist control (No Intervention): Participants of the waitlist control group will not receive any training while the other three group are having their interventions. After the completion of the all assessments, the participants will receive the 12-week qigong training, same as the qigong group.

INTERVENTIONS:
Behavioral: Qigong (Baduanjin) — Participants will receive 24 sessions of Baduanjin training over 12 weeks (2 sessions per week). Each session will last for 60 minutes. Baduanjin consists of eight forms of gentle movements, and it takes about 10 to 15 minutes to complete a full cycle. Participants will learn to practice each form gradually over the first 12 sessions. In the remaining 12 sessions, the participants will go through all the movements 2-3 times, with guided practice on rhythmic breathing and mind regulation (attention to body and breathing) to be performed in coordination with the movements. The training will be delivered by an instructor after training by the project team.
  Arms: Qigong (Baduanjin)
Behavioral: Mindfulness-based intervention — Participants will receive mindfulness-based intervention with the same duration and frequency as qigong group. The intervention incorporates psychoeducation on mindfulness and stress management and group-based mindfulness practice about breathing, awareness of body sensations, thoughts, stretching, and walking. All the mindfulness practices are based on publicly accessible audio recordings. The training will be delivered by an instructor after training by the project team.
  Arms: Mindfulness-based intervention
Behavioral: Physical exercise — Participants of the physical exercise group will receive training of a series of low-to-moderate intensity physical activities for the same duration and frequency as qigong group. The physical activities include stretching, flexibility exercise, balance exercise, and aerobic exercise. The training will be delivered by an instructor after training by the project team.
  Arms: Physical exercise

SUMMARY:
One goal of the study is to evaluate the efficacy of qigong to alleviate depressive symptoms and enhance cognitive function in comparison to mindfulness-based intervention, physical exercise, and waitlist control. The other goal is to explore the changes in neurobiological markers that may explain the qigong-related effects on depressive symptoms and cognitive function. The main research questions are:

* Is the 12-week qigong training more effective than mindfulness-based intervention, physical exercise, and waitlist control to alleviate depressive symptoms?
* Is the 12-week qigong training more effective than mindfulness-based intervention, physical exercise, and waitlist control to enhance cognitive function?

Participants are older adults aged 60 or above. They were randomly assigned to qigong training, mindfulness training, physical exercise training, or wait-list which all last for 12 weeks. Their changes before and after the 12-week period in depressive symptoms, neurobiological markers, and cognitive functions are assessed.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older;
* With mild or severer levels of depressive symptoms as indicated by the Geriatric Depression Scale (GDS-8) scores of 5 or above, or Depression Anxiety and Stress Scale-21 (DASS-21) depression subscale scores of 4 or above
* Self-identified as physically stable and without life-threatening diseases.
* Be able to communicate in Cantonese or Mandarin.

Exclusion Criteria:

* Have a history of practicing or receiving training of any form of mind-body or regular exercises (including tai chi, yoga, and qigong, or regular physical activity > 3 times/week) during the month prior to intervention
* Have changed medications or the dose of medications prescribed for their health condition in the one month prior to study enrollment
* Have severe cognitive or language impairment based on the assessment with Montreal Cognitive Assessment (MoCA)
* Taking medication or undergoing electroconvulsive therapy, psychotherapy, or psychoeducation for a psychological or psychiatric condition
* Unable to demonstrate satisfactory standing balance

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline and post-intervention (12 weeks after baseline)
  The eight-item Patient Health Questionnaire
Global cognitive function | Baseline and post-intervention (12 weeks after baseline)
  Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Serum adiponectin | Baseline and post-intervention (12 weeks after baseline)
  Collected and assayed through peripheral blood sample
Serum BDNF | Baseline and post-intervention (12 weeks after baseline)
  Collected and assayed through peripheral blood sample
Salivary cortisol | Baseline and post-intervention (12 weeks after baseline)
  Collected and assayed through saliva sample
Attention | Baseline and post-intervention (12 weeks after baseline)
  Attention Network Task
Inhibitory control | Baseline and post-intervention (12 weeks after baseline)
  Attention Network Task
Working memory | Baseline and post-intervention (12 weeks after baseline)
  N-back Task
ERP N2 amplitude | Baseline and post-intervention (12 weeks after baseline)
  ERP data recorded during Attention Network Task and N-back Task
ERP P3 amplitude | Baseline and post-intervention (12 weeks after baseline)
  ERP data recorded during Attention Network Task and N-back Task
Hand grip strength | Baseline and post-intervention (12 weeks after baseline)
  To be assessed with a Jamar handheld dynamometer
Affect | Baseline and post-intervention (12 weeks after baseline)
  Positive and Negative Affect Schedule

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Department of Rehabilitation Sciences, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No